CLINICAL TRIAL: NCT01062022
Title: FOCUS-CI: A Preventive Intervention With Children and Families of the Combat Injured
Acronym: FOCUS-CI
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Loss of funding
Sponsor: Henry M. Jackson Foundation for the Advancement of Military Medicine (Other)
Collaborators: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: G188NI; W81XWH-08-2-0650 (Other Grant/Funding Number: CDMRP)
Record Dates: First submitted 2010-02-01; First posted 2010-02-04 (Estimated); Last update posted 2016-08-18 (Estimated); Status verified 2016-08

CONDITIONS: Stress Disorders; Combat Disorders; Traumatic Stress Disorders
Keywords: intervention; combat wounded; family; Focus-CI
MeSH Terms: conditions — Stress Disorders, Traumatic; Combat Disorders | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control - Standard of Care (Active Comparator): Participation in the study will involve your child completing a questionnaire about (a) your family's background, descriptive information about people in your family, and previous major life events, (b) his/her current functioning, (c) his/her feelings before, during, and after the combat injury, and (d) his/her current social relationships and adjustment. Your child will be asked to complete the questionnaire during the baseline assessment, and at 6 months, 12 months, and 24 months after the original assessment.
  Interventions: Behavioral: Standard of Care
- FOCUS-CI (Active Comparator): Those participants in the FOCUS-CI intervention will be part of a family skill-building/resiliency training program designed to provide information and skills training in a variety of forms, including clinician-led sessions, handouts, on-line training modules, and individual family care management. Study participation will also involve completing a questionnaire about (a) your family's background, descriptive information about people in your family, and previous major life events, (b) his/her current functioning, (c) his/her feelings before, during, and after the combat injury, and (d) his/her current social relationships and adjustment. Questionnaires will be completed during the baseline assessment, and at 6 months, 12 months, and 24 months after the baseline assessment.
  Interventions: Behavioral: FOCUS-CI

INTERVENTIONS:
Behavioral: Standard of Care — Families randomized to this arm will receive the standard of care. They will be compared to the families in the FOCUS-CI arm of the study.
  Other Names: comparison group, standard of care
  Arms: Control - Standard of Care
Behavioral: FOCUS-CI — Families randomized to this arm of the study will be part of a family skill-building/resiliency training program designed to provide information and skills training
  Other Names: FOCUS-CI, Families OverComing Under Stress-Combat Injury
  Arms: FOCUS-CI

SUMMARY:
The purpose of this study is to implement a unique evidence-based intervention program to help military families deal with the critical issue of combat injury and its impact on current and future family health and functioning. The study is a randomized study. The study will compare the effects of the newly designed FOCUS-CI (Families OverComing Under Stress - Combat Injury) with the existing standard of care (SoC) at three military medical rehabilitation sites (Walter Reed Amry Medical Center, Brooke Army Medical Center and Madigan Army Medical Center) on key aspects of family health and functioning.

DETAILED DESCRIPTION:
Injured service members who have at least one child between the ages of 5 and 18 years who have sustained a combat injury severe enough to require at least two weeks of inpatient hospitalization and who are within 6 months of discharge from inpatient hospitalization and currently receiving outpatient care will be recruited into this study.

ELIGIBILITY:
Inclusion Criteria:

For a family to be eligible for the study, the injured service member must:

* have sustained a combat injury that was severe enough to require a minimum of two weeks inpatient hospitalization immediately after the injury;
* currently be participating in outpatient rehabilitation for the same combat injury;
* must be within 6 months of discharge from inpatient hospitalization at the start of the intervention;
* families must have at least one child between the ages of 5 and 18 and be fluent in English. English fluency will be determined by asking, "Is English spoken in your home?"
* pregnant women are eligible to participate.

Exclusion Criteria:

* families in which the service member did not sustain a qualifying injury or has been discharged from inpatient care for more than six months will not be eligible to participate
* families in which a member is actively psychotic
* families in which a service member's primary relationship is with a "significant other" who is not eligible for military medical care
* due to the limited ability of young children to comprehend the intervention activities, children under the age of 5 years will not be invited to participate in the intervention.
* no one will be excluded based on race, ethnicity, gender, pregnancy, medical status, or cognitive functioning.

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2011-01; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
parent and child distress (including mental health service usage, symptoms of PTSD and Depression) | every 12 months

SECONDARY OUTCOMES:
Participant Satisfaction with Intervention | every 12 months
Clinician Satisfaction with Intervention | months 12 and 24 at followup
Parent Functioning (including substance use, parental efficacy, parental satisfaction, parenting behavior, social support and posttraumatic growth) | at 12 and 24 month followups
Child Functioning (School Functioning, and Coping) Family Functioning (Communication, Problem Solving, Roles, and Relationships) | at 12 and 24 month followup

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Cozza, MD, Principal Investigator — Uniformed Services University of the Health Sciences (USUHS); Robert Ursano, MD, Study Chair — Uniformed Services University of the Health Sciences (USUHS)
Locations (3):
- United States (3):
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - Brooke Army Medical Center, San Antonio, Texas
  - Madigan Army Medical Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Undecided
study ended - no data

REFERENCES:
- See also: USUHS — http://www.usuhs.edu
- See also: Henry M. Jackson Foundation for the Advancement of Military Medicine — http://www.hjf.org